CLINICAL TRIAL: NCT06857318
Title: Colostrum From MERS-CoV Seropositive Camels for SARS-CoV-2 Infection - From Lab to Human- a Placebo Controlled Randomized Trial.
Brief Title: Colostrum From MERS-CoV Seropositive Camels for SARS-CoV-2 Infection - a Placebo-controlled Randomized Trial.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Hila Elinav, Director of Hadassah AIDS center, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMO-238-20
Record Dates: First submitted 2025-02-27; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: COVID 19
Keywords: infectivity; viral load; MERS-Cov; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Water; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colostrum Treatment Group (Experimental)
  Interventions: Biological: Colostrum Nasal Spray
- Control (Placebo Comparator)
  Interventions: Other: Water for injection

INTERVENTIONS:
Biological: Colostrum Nasal Spray — 24 hours use of nasal spray of colostrum from MERS-CoV positive camels- 6 doses total
  Arms: Colostrum Treatment Group
Other: Water for injection — 24 hours use of a nasal spray of water for injection- 6 doses total
  Arms: Control

SUMMARY:
The study aims to study the efficacy of colostrum from MERS-CoV-positive camels applied as a nasal spray to COVID-19 patients for treatment and prevention of SARS-CoV-2 infection. This study will compare the usage of colostrum to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Laboratory-proven infection with COVID-19 using PCR or another approved kit
* Hospitalized / community setting-at low-moderate clinical risk according to the NEWS-2 scale with a score of 0-10.
* Onset of symptoms up to 7 days before inclusion
* Can sign informed consent
* Willingness and ability to participate in research

Exclusion Criteria:

* Pregnant women or lactating
* Lack of judgment (psychiatric disorder or dementia)
* Immunosuppressed - HIV with CD4 below 500, chemotherapy, steroids - more than 5 mg per day, solid organ transplants, bone marrow transplants, active hematological or oncological malignancies, biological therapy
* Neutropenia (less than 2000 neutrophils per cubic meter) or thrombocytopenia (platelet count less than 50000 per cubic meter).
* Acute or chronic sinusitis.
* Nasal polyps or any pathology in the nasal cavity
* Cystic fibrosis
* Significant disturbance in liver functions (AST/ALT more than 5 times the ULN)
* Significant renal dysfunction (GFR lower than 30 ml per minute)
* Known allergy to colostrum or cow's milk
* Use of another study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Viral Load and Infectivity | 24 hours
  Viral load and infectivity will be measured using nasal swabs

SECONDARY OUTCOMES:
Undetectable Viral Load and Non-infectious Virus | 72 hours
  Viral load and infectious virus will be assessed by nasal swabs

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Hebrew University, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided